CLINICAL TRIAL: NCT04046913
Title: The ADDapt Diet in Reducing Crohn's Disease Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRAS 260196
Record Dates: First submitted 2019-07-26; First posted 2019-08-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases
Keywords: Dietary intervention
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low food additive diet (Active Comparator): Dietary advice, given by a dietitian, will be discussed at trial baseline.
  Interventions: Behavioral: Dietary education
- Habitual food additive diet (Placebo Comparator): Dietary advice, given by a dietitian, will be discussed at trial baseline.
  Interventions: Behavioral: Dietary education

INTERVENTIONS:
Behavioral: Dietary education — Intervention: Low food additive diet. Control: Habitual food additive diet

SUMMARY:
Crohn's disease (CD) results in chronic intestinal inflammation, is of increasing incidence both in the developed and developing world and has a marked impact on patient quality of life. The prevalence of CD is 10.6 per 100,000 people in the UK and represents a significant annual financial burden of around €16.7 billion in Europe.

A wide range of nutrients and food components have been investigated for their role in the pathogenesis and course of CD. A common theme suggests that CD risk is associated with a "Western diet", including high fat, high sugar and processed foods. However, intervention studies that exclude specific aspects of the diet such as sugar or that compare low and high fat diets have failed to show effectiveness in practice. Observational human and experimental animal studies suggest that certain food additives used extensively by the food industry play a role in the pathogenesis and natural history of CD. However, to date no evidence exists for the effectiveness of a diet low in these food additives in CD.

Therefore, the aim of this study is to investigate the effects of a diet low in certain food additives compared to a normal UK diet on CD activity, health-related quality of life, gut bacteria, gut permeability, gut inflammation and dietary intake, in patients with mildly active, stable CD. We will recruit patients with mildly active CD and will randomise them to receive either the diet low in the food additives of interest, or the diet representative of a normal UK diet. Patients will follow their allocation diet for 8 weeks and will attend study visits at the start and end of the trial, at which points questionnaires will be completed and samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥16 years
* CD diagnosis (defined by standard clinical, histological and radiological criteria) of at least 3 months
* Mildly active disease as defined by:

  * Defined by physician assessment that no change in medication is required
  * Faecal calprotectin >150 µg/g OR endoscopic evidence of active luminal disease OR radiological evidence of active luminal disease (by magnetic resonance enterography, or ultrasound) within the last 8 weeks.
  * CDAI between 150-250
* Current body weight of ≥50 kg
* Individuals able to give informed consent and willingness to participate

Exclusion Criteria:

* Changes in dose to azathioprine, 6-mercaptopurine, methotrexate or anti-TNF-α agents or other biologics during the preceding 8 weeks, oral 5-ASA during the preceding four weeks. Currently receiving oral prednisolone/budesonide or discontinued within the last 4 weeks, unless they are on a stable dose of 10 mg/day or less prednisolone (3 mg or less budesonide) for at least 4 weeks with the intention to continue this long term.
* Used rectal 5-ASA or rectal steroids in the preceding 4 weeks
* Previous extensive bowel resection, defined as having had >2 intestinal resections, a sub-total colectomy or documented short bowel syndrome
* Poorly controlled bile acid malabsorption
* Current stoma
* Recent use of the following treatments: antibiotics, probiotics, prebiotic or fibre supplements in the preceding four weeks, NSAIDs during the preceding week
* Full bowel preparation for a diagnostic procedure in preceding 4 weeks
* Comorbidities including sepsis/fever, diabetes or coeliac disease, or other concomitant serious comorbidity e.g. significant psychiatric, hepatic, renal, endocrine, respiratory, neurological or cardiovascular disease
* Exclusive enteral nutrition in the past 8 weeks
* Assessed as at nutritional risk, as defined by any of the following:

  * BMI ≤18.5 kg/m2
  * Previous or current eating disorder
  * Currently receiving prescribed oral nutritional supplements
* Following a restrictive diet (e.g. multiple restrictions due to numerous self-reported allergies) as judged by the dietitian
* Reported pregnancy or lactation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index | Difference between baseline and week 8
  The proportion of patients achieving at least a 70-point reduction in the Crohn's Disease Activity Index from baseline to week 8

SECONDARY OUTCOMES:
Faecal calprotectin | Baseline, 8 weeks and 26 weeks
  The proportion of patients achieving at least a 50% reduction in faecal calprotectin concentration.
Faecal calprotectin | Baseline, 8 weeks and 26 weeks
  Absolute and change in faecal calprotectin concentrations during the trial.
Faecal calprotectin | Baseline, 8 weeks and 26 weeks
  Proportion of patients achieving faecal calprotectin concentrations <150 µg/g.
Serum C-reactive protein | Baseline, 8 weeks and 26 weeks
  Absolute and change in CRP concentration and proportion of patients achieving a CRP concentration <5 mg/L
Mucosal immune cell gene expression | Baseline and 8 weeks
  RNA sequencing on GI immune cells isolated from rectal biopsies
Crohn's Disease Activity Index (CDAI) | Baseline, 8 weeks and 26 weeks
  Absolute and change in CDAI score during the trial.
Crohn's Disease Activity Index (CDAI) | Baseline and 8 weeks
  Proportion of patients achieving a CDAI score <150 points (clinical remission) by 8 weeks.
Crohn's Disease Activity Index (CDAI) | Baseline and 8 weeks
  Proportion of patients achieving ≥100-point reduction in CDAI score by 8 weeks.
Stool Output | Baseline, 8 weeks and 26 weeks
  Absolute and change in stool frequency and consistency
Perceived Crohn's disease control | Baseline, 8 weeks and 26 weeks
  Absolute and change in score in IBD-control questionnaire
Health related quality of life | Baseline, 8 weeks and 26 weeks
  Absolute and change in Inflammatory Bowel Disease questionnaire (IBDQ) score, and proportion of patients achieving clinical remission i.e., IBDQ score >168
Faecal microbiota composition | Baseline, 8 weeks and 26 weeks
  Shotgun sequencing
Faecal microbial gene expression | Baseline, 8 weeks and 26 weeks (in a subset of participants)
  Meta-transcriptomics
Mucosal microbiota composition | Baseline and 8 weeks (in a subset of participants)
  16S sequencing
Gastrointestinal permeability | Baseline and 8 weeks
  Sugar probe solution urinary analysis to determine intestinal permeability
Dietary intake | Baseline, 8 weeks and 26 weeks
  Micronutrient and macronutrient intake, food intake and dietary pattern
Dietary adherence | Baseline, 8 weeks and 26 weeks
  Reduction in intake of food additives and consumption of study foods and snacks
Diet feasibility and acceptability | Baseline, 8 weeks and 26 weeks
  Acceptability questionnaire, including food-related quality of life
Physical Activity | Baseline, 8 weeks and 26 weeks
  International Physical Activity Questionnaire
Metabolomics | Baseline and 8 weeks
  Metabolomics analyses through Liquid Chromatography - Mass Spectrometry using validated assays.
Biomarker study | Baseline and 8 weeks
  Biomarker study through Nuclear Magnetic Resonance Spectroscopy
Genetics | Baseline
  Whole genome single nucleotide polymorphism array genotyping

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided